CLINICAL TRIAL: NCT00571064
Title: A 12-Week, Multicenter, Open Label Study To Evaluate The Effectiveness And Safety Of Donepezil Hydrochloride (E2020) In Subjects With Mild To Severe Alzheimer's Disease Residing In An Assisted Living Facility
Brief Title: The Effectiveness And Safety Of Donepezil Hydrochloride (E2020) In Subjects With Mild To Severe Alzheimer's Disease Residing In An Assisted Living Facility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2020-A001-415
Record Dates: First submitted 2007-12-06; First posted 2007-12-11 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-02

CONDITIONS: Mild to Severe Alzheimer's Disease
MeSH Terms: interventions — Donepezil

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Donepezil HCl

INTERVENTIONS:
Drug: Donepezil HCl — One 5 mg tablet per day (for the first 6 weeks) with a full glass of water. For the last 6 weeks, one 10mg tablet per day with a full glass of water.
  Other Names: Aricept

SUMMARY:
This is a study to determine the effectiveness and safety of donepezil hydrochloride (E2020) used to treat residents of assisted living facilities diagnosed with mild, moderate, or severe stage Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: Subjects > 50 years of age.
2. Sex distribution: both men and women. Women must be two (2) years post-menopausal or surgically sterile. Women of child bearing potential (< 1 year post menopausal) must be practicing effective contraception and have a negative ß-hCG at screening (Women who are breast feeding are excluded).
3. MMSE scores between 5 and 24 (inclusive).
4. Subjects must have diagnostic evidence of possible or probable AD either prior to or at the screening visit based on Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) and National Institute of Neurological and Communicative Disorders and Stroke criteria.
5. CT or MRI within the last 12 months consistent with a diagnosis of AD without any other clinically significant comorbid pathologies found. A copy of the report will be required and will be collected. If there has been a significant change in clinical status suggestive of stroke or other neurological disease in addition to AD with onset between the time of the last CT or MRI and the screening evaluation, the scan should be repeated during screening.
6. The caregiver/ informant can be a family member or a professional and must have had contact with the subject at least 6 Weeks prior to study entry and spent at minimum 3 days a Week (10 hours per Week) with the subject. For study visit, the subject can be seen at the Assisted Living Facility (ALF) or in the clinic setting of the Investigator. At each visit, the caregiver/informant will provide the information for completion of the safety and efficacy assessments based on knowledge of and time spent with the subject.
7. Subjects must reside in an ALF.
8. The subject is expected to complete all procedures scheduled during the screening, baseline, interim, and final visits including all efficacy assessments.
9. Putative non-prescription/prescription cognitive enhancers (e.g. ginkgo, high-dose vitamin E, lecithin, estrogen, non-steroidal anti-inflammatory drugs [NSAIDs]) will not be excluded but will be discouraged. If a putative cognitive enhancer is present, the dosage must have been stable for at least 3 months prior to the screening visit and should not change during the course of the study.
10. Subjects with controlled hypertension (sitting diastolic BP < 95 mmHg), right bundle branch block (complete or partial), and pacemakers may be included in the study.
11. Subjects with thyroid disease also may be included in the study provided they are euthyroid and stable on treatment for at least 3 months prior to screening.
12. Subjects with a history of seizure disorder are allowed provided that they are on stable treatment for at least 3 months prior to screening and have not had a seizure within the past 6 months.
13. Subjects must be able to swallow tablet medication -- no crushing of tablet is allowed.
14. Health: independent or ambulatory aided (i.e., walker or cane, to wheelchair); vision and hearing (eyeglasses and/or hearing aid permissible) sufficient for compliance with testing procedures.
15. Subjects must be sufficiently proficient in the language in which the assessments are to be conducted.
16. Subjects must have clinical laboratory values within normal limits, and within the Eisai (sponsor) guidelines, or abnormalities considered not clinically significant by the investigator and sponsor.

Exclusion Criteria:

1. Age range: Subjects < 50 years of age.
2. MMSE score of ≤4 or ≥25.
3. Subjects with active or clinically significant conditions affecting absorption, distribution or metabolism of the study medication (e.g., inflammatory bowel disease, gastric or duodenal ulcers or severe lactose intolerance).
4. Subjects with a known hypersensitivity to piperidine derivatives or cholinesterase inhibitors.
5. Subjects living in a skilled nursing home or subjects living in an ALF who may be moved to a skilled nursing home during the course of the study. Subjects who transfer from an ALF to a skilled nursing home during this study will be discontinued.
6. Subjects who have taken the following medications within the last 3 months prior to screening will be not eligible: Aricept, Exelon, Cognex, Razadyne, Metrifonate, Namenda or propentofylline.
7. Subjects without a reliable caregiver/informant or subjects whose caregiver is unwilling or unable to complete the outcome measures and fulfill the requirements of this study.
8. Subjects with clinically significant obstructive pulmonary disease or asthma, untreated for > 3 months.
9. Subjects with recent (< 2 years) hematologic/ oncologic disorders, not including mild anemia or basal or squamous cell carcinoma of the skin. Subjects with current evidence of malignant neoplasm or recurrent or metastatic disease will be excluded.
10. Evidence of clinically significant, active gastrointestinal, renal, hepatic, endocrine or cardiovascular system disease.
11. Subject with a current DSM-lV diagnosis of Major Depressive Disorder (MDD) or any current primary psychiatric diagnosis other than Alzheimer's disease (as per DSM-lV).
12. Subjects with dementia complicated by other organic disease (DSM 290.30 or 290.11) are excluded; depression or delusions are common in Alzheimer's disease, and subjects with severe symptoms so pronounced that they warrant an alternative, concurrent diagnosis, are excluded.
13. Subjects with a known or suspected history of alcoholism or drug abuse (within the past 10 years).
14. Subjects with treated hypothyroidism that have not been on a stable dose of medication for 3 months prior to screening and who do not have normal serum Free T3, Free T4 and TSH at screening.
15. Subjects with treated vitamin B-12 deficiency who have not been on a stable dose of medication for at least 3 months prior to the study screening visit and who do not have normal serum B-12 levels at screening.
16. Any subject taking a prohibited medication will be excluded.
17. Any condition which would make the subject or the caregiver, in the opinion of the investigator, unsuitable for the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2009-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Prodafikas, MD, Study Director — Eisai Inc.
Locations (36):
- United States (36):
  - Senior Care, Birmingham, Alabama
  - 21st Century Neurology, Phoenix, Arizona
  - Psypharma Clinical Research, Phoenix, Arizona
  - South Coast Clinical Trials, Anaheim, California
  - AVI Clinical Research, Carson, California
  - Margolin Brain Institute, Fresno, California
  - Sarah Sam Olelewe, MD Inc, Hawthorne, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Danbury Clinical Research, LLC, Danbury, Connecticut
  - Research Center for Clinical Studies, Norwalk, Connecticut
  - Neuroscience Consultants, Miami, Florida
  - Galiz Research, Miami Springs, Florida
  - Universal Clinical research and Technology, Orlando, Florida
  - Byrd's Alzheimer Institute, Tampa, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Center for Clinical Trials, Venice, Florida
  - Rush Alzheimer Disease Center, Chicago, Illinois
  - Alexian Brothers Neuroscience Institute, Elk Grove, Illinois
  - Agewell Health Ltd, Indianapolis, Indiana
  - Venture Resource Group Inc, Mission, Kansas
  - Four Rivers Clinical Research, Paducah, Kentucky
  - McLean Hospital Geriatric Psychiatry, Belmont, Massachusetts
  - Neuroscience Research of the Bershires, Pittsfield, Massachusetts
  - Horne Research, Las Vegas, Nevada
  - Bio Behavioral Health, Toms River, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Neurological Associates of Albany, PC, Albany, New York
  - University Of Buffalo, Buffalo, New York
  - University of Rochester, Monroe Community Hospital, Rochester, New York
  - Valley Medical Research, Centerville, Ohio
  - Infinity Research Group, Oklahoma City, Oklahoma
  - University of Pennsylvania, Section of Geriatric Psychiatry, Philadelphia, Pennsylvania
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - CNS Research, INC, East Providence, Rhode Island
  - Senior Adults Specialty Research, Austin, Texas
  - Mech Center, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil Hydrochloride (HCl): Donepezil HCl 5 milligrams (mg) per day (one 5 mg tablet) was administered for the first 6 weeks (42 days), and then the dose was increased to 10 mg/day (two 5 mg tablets). If 10 mg of donepezil was not tolerated, the dosage was reduced temporarily to 5 mg. The participant was re-challenged with 10 mg of study drug within 5 to 7 days. If the participant still could not tolerate the higher dose after re-challenge, they continued in the study on 5 mg per day of study drug.
Period: Overall Study
Arm/Group | Donepezil Hydrochloride (HCl)
Started | 97
Completed | 76
Not Completed | 21
Not completed — Adverse Event | 13
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who took at least one dose of study medication.
Groups:
- Donepezil Hydrochloride (HCl): Donepezil HCl 5 milligram (mg) per day (one 5 mg tablet) was administered for the first 6 weeks (42 days), and then the dose was increased to 10 mg/day (two 5 mg tablets). If 10 mg of donepezil was not tolerated, the dosage was reduced temporarily to 5 mg. The participant was re-challenged with 10 mg of study drug within 5 to 7 days. If the participant still could not tolerate the higher dose after re-challenge, they continued in the study on 5 mg per day of study drug.
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 81.0 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Mini Mental State Examination (MMSE) Total Scores by Visit
Description: The MMSE was a brief test that assessed the cognitive status of the participant. The 30-point test included items that evaluate orientation to time and place, immediate and delayed recall, attention, language, and construction. The total number of correct responses was obtained. The scores ranged from 0 to 30, with higher scores representing better performance. Summaries and analyses in the Intent-to-Treat (ITT) population were carried out using observed cases at each visit. A Study Endpoint evaluation was performed using the last observation carried forward (LOCF) from the open label treatment phase for each participant. The outcome of the study was based on analyses of the primary efficacy variable at Study Endpoint, which was defined as end of study assessment, using the ITT population with LOCF.
Time Frame: Baseline (Visit 2), Week 6 (Visit 3), Week 12 (Visit 4) or Early Termination (ET) Visit, Week 12 LOCF (Study Endpoint)
Population: ITT population with LOCF included all enrolled participants who took at least one dose of study medication, and had baseline and at least one post-baseline assessment of at least one efficacy variable.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 93
Scores on a scale
  Baseline (Visit 2) | 18.7 (5.29)
  Week 6 (Visit 3) | 20.8 (5.16)
  Week 12/ET (Visit 4) | 20.5 (5.92)
  Week 12 LOCF (Study Endpoint) | 20.5 (5.88)

2. Secondary Outcome: Caregiver Activity Survey (CAS) Total Time by Visit
Description: The CAS was a validated tool that measured the time caregivers spent aiding Alzheimer's participants with their day-to-day activities. The CAS recorded time spent on six activities of daily living, communicating with the person, using transportation, dressing, eating, looking after one's appearance, and supervising the person. Caregivers were asked to report the amount of time spent on each activity during a 'typical' caregiving day. Total time for the CAS was calculated as the sum of the sub-item times.
Time Frame: Baseline (Visit 2), Week 6 (Visit 3), Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint)
Population: ITT population included all enrolled participants who took at least one dose of study medication, and had baseline and at least one post-baseline assessment of at least one efficacy variable. Study endpoint evaluation at week 12 included ITT population with LOCF.
Measure: Mean (Standard Deviation); unit: Hours/day
Groups:
- Donepezil Hydrochloride (HCl): Donepezil HCl 5 mg per day (one 5 mg tablet) was administered for the first 6 weeks (42 days), and then the dose was increased to 10 mg/day (two 5 mg tablets). If 10 mg of donepezil was not tolerated, the dosage was reduced temporarily to 5 mg. The participant was re-challenged with 10 mg of study drug within 5 to 7 days. If the participant still could not tolerate the higher dose after re-challenge, they continued in the study on 5 mg per day of study drug.
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 93
Hours/day
  Baseline (Visit 2) | 8.9 (8.80)
  Week 6 (Visit 3) | 9.0 (9.99)
  Week 12/ET (Visit 4) | 9.0 (9.81)
  Week 12 LOCF (Study Endpoint) | 9.3 (10.07)

3. Secondary Outcome: Change From Baseline in CAS Total Time by Visit
Description: The CAS was a validated tool that measured the time caregivers spent aiding Alzheimer's participants with their day-to-day activities. The CAS recorded time spent on six activities of daily living, communicating with the person, using transportation, dressing, eating, looking after one's appearance, and supervising the person. Caregivers were asked to report the amount of time spent on each activity during a 'typical' caregiving day. Total time for the CAS was calculated as the sum of the sub-item times. Change from Baseline in CAS Total Time at Week 6 (Visit 3), Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint) has been reported.
Time Frame: Baseline, Week 6 (Visit 3), Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours/day
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 93
Hours/day
  Baseline | 8.9 (8.80)
  Change from Baseline at Week 6 (Visit 3) | 0.3 (6.83)
  Change from Baseline at Week 12/ET (Visit 4) | 0.3 (5.82)
  Change from Baseline at Week 12 LOCF | 0.3 (5.78)
Statistical Analysis 1: Comparison: Donepezil Hydrochloride (HCl); Week 6 (Visit 3); Test type: Superiority or Other; p = 0.6593, t-test, 2 sided — Significance level of 0.05
Statistical Analysis 2: Comparison: Donepezil Hydrochloride (HCl); Week 12/ET (Visit 4); Test type: Superiority or Other; p = 0.6048, t-test, 2 sided — Significance level of 0.05
Statistical Analysis 3: Comparison: Donepezil Hydrochloride (HCl); Week 12 LOCF (Study Endpoint); Test type: Superiority or Other; p = 0.5924, t-test, 2 sided — Significance level of 0.05

4. Primary Outcome: Change From Baseline in MMSE Total Score by Visit
Description: The MMSE was a brief test that assessed the cognitive status of the participant. The 30-point test included items that evaluated orientation to time and place, immediate and delayed recall, attention, language, and construction. The total number of correct responses was obtained. The scores ranged from 0 to 30, with higher scores representing better performance. Summaries and analyses in the ITT population were carried out using observed cases at each visit. A Study Endpoint evaluation was performed using the LOCF from the open label treatment phase for each participant. The outcome of the study was based on analyses of the primary efficacy variable at Study Endpoint, which was defined as end of study assessment, using the ITT population with LOCF. Change from Baseline in MMSE Total Score at Week 6 (Visit 3), Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint) has been reported.
Time Frame: Baseline, Week 6 (Visit 3), Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 93
Scores on a scale
  Baseline | 18.7 (5.29)
  Change from Baseline at Week 6 (Visit 3) | 1.8 (2.81)
  Change from Baseline at Week 12/ET (Visit 4) | 1.9 (2.79)
  Change from Baseline at Week 12 LOCF | 1.8 (2.81)
Statistical Analysis 1: Comparison: Donepezil Hydrochloride (HCl); Week 6 (Visit 3); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Significance level 0.05
Statistical Analysis 2: Comparison: Donepezil Hydrochloride (HCl); Week 12/ET (Visit 4); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Significance level of 0.05
Statistical Analysis 3: Comparison: Donepezil Hydrochloride (HCl); Week 12 LOCF (Study Endpoint); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Significance level of 0.05

5. Secondary Outcome: Neuropsychiatric Inventory (NPI-8) Total Score by Visit
Description: The NPI-8 was an 8-item scale that assessed eight behavioral domains: delusions, hallucinations, agitation, depression, anxiety, apathy, irritability, and aberrant motor behavior. The frequency (0 to 4) and severity (0 to 3) of each domain were assessed; the sub-score for each domain was calculated as the product of the frequency and severity rating. The total score for the NPI was calculated as the sum of the domain sub-score, range from 0 to 96, with higher scores indicating greater behavior disturbances.
Time Frame: Baseline (Visit 2), Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 93
Scores on a scale
  Visit 2 (Baseline) | 5.7 (9.70)
  Week 12/ET (Visit 4) | 3.9 (5.73)
  Week 12 LOCF (Study Endpoint) | 3.9 (5.73)

6. Secondary Outcome: Change From Baseline in NPI-8 Total Score by Visit
Description: The NPI-8 was an 8-item scale that assessed eight behavioral domains: delusions, hallucinations, agitation, depression, anxiety, apathy, irritability, and aberrant motor behavior. The frequency (0 to 4) and severity (0 to 3) of each domain were assessed; the sub-score for each domain was calculated as the product of the frequency and severity rating. The total score for the NPI was calculated as the sum of the domain sub-score, range from 0 to 96, with higher scores indicating greater behavior disturbances. Change from Baseline in NPI-8 Total Score at Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint) has been reported.
Time Frame: Baseline, Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 93
Scores on a scale
  Baseline | 5.7 (9.7)
  Change from Baseline at Week 12/ET (Visit 4) | -1.8 (8.39)
  Change from Baseline at Week 12 LOCF | -1.8 (8.39)
Statistical Analysis 1: Comparison: Donepezil Hydrochloride (HCl); Week 12/ET (Visit 4); Test type: Superiority or Other; p = 0.0431, t-test, 2 sided — Significance level of 0.05
Statistical Analysis 2: Comparison: Donepezil Hydrochloride (HCl); Week 12 LOCF (Study Endpoint); Test type: Superiority or Other; p = 0.0431, t-test, 2 sided — Significance level of 0.05

7. Secondary Outcome: Alzheimer Disease-related Quality of Life (ADRQL) Total Score by Visit
Description: The ADRQL was an observer-rated quality of life instrument that measured the following domains: social interaction, awareness of self, feelings and mood, enjoyment of activities, and response to surroundings. The ADRQL was a 47-item questionnaire with five domains: relating to and being around other people (ADRQL-A; 12 items), a person's special identity and important relationships (ADRQL-B; 8 items), different types of behavior (ADRQL-C; 15 items), usual activities (ADRQL-D; 5 items), and behavior in a person's living environment (ADRQL-E; 7 items). Domain sub-scores were summed to yield a total raw score, which was divided by the total possible score and multiplied by 100 to produce the final score. Each subscale score could be calculated in the similar approach. Total score ranges from 0-100 where higher scores reflected a better quality of life.
Time Frame: Baseline (Visit 2), Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 93
Scores on a scale
  Baseline (Visit 2) | 48.7 (8.71)
  Week 12/ET (Visit 4) | 47.6 (7.90)
  Week 12 LOCF (Study Endpoint) | 47.6 (7.90)

8. Secondary Outcome: Change From Baseline in ADRQL Total Score by Visit
Description: The ADRQL was an observer-rated quality of life instrument that measured the following domains: social interaction, awareness of self, feelings and mood, enjoyment of activities, and response to surroundings. The ADRQL was a 47-item questionnaire with five domains: relating to and being around other people (ADRQL-A; 12 items), a person's special identity and important relationships (ADRQL-B; 8 items), different types of behavior (ADRQL-C; 15 items), usual activities (ADRQL-D; 5 items), and behavior in a person's living environment (ADRQL-E; 7 items). Domain sub-scores were summed to yield a total raw score, which was divided by the total possible score and multiplied by 100 to produce the final score. Each subscale score could be calculated in the similar approach. Higher scores reflected a better quality of life. Change from Baseline in ADRQL Total Score at Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint) has been reported.
Time Frame: Baseline, Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 93
Scores on a scale
  Baseline | 48.7 (8.71)
  Change from Baseline at Week 12/ET (Visit 4) | -1.1 (6.93)
  Change from Baseline at Week 12 LOCF | -1.1 (6.93)
Statistical Analysis 1: Comparison: Donepezil Hydrochloride (HCl); Week 12/ET (Visit 4); Test type: Superiority or Other; p = 0.1285, t-test, 2 sided — Significance level of 0.05
Statistical Analysis 2: Comparison: Donepezil Hydrochloride (HCl); Week 12 LOCF (Study Endpoint); Test type: Superiority or Other; p = 0.1285, t-test, 2 sided — Significance level of 0.05

9. Secondary Outcome: Disability Assessment in Dementia (DAD) Total Score by Visit
Description: The DAD was a 10 domain 40-item scale that measured a participant's ability to initiate, plan, organize, and perform both basic and instrumental activities of daily living. These domains were: hygiene (7 items), dressing (5 items), continence (2 items), eating (3 items), meal preparation (3 items), telephoning (4 items), going on an outing (5 items), finance (4 items), medication (2 items), and leisure (5 items). The three responses to the DAD items were "No, Yes, and N/A". A "No" answer scored 0 and a "Yes" answer scored 1. The scoring range was 0-40, with a higher score indicating less disability (better quality of life). If N/A was selected then it was treated as missing. When there were items with missing values, the domain sub-scores and the total score were imputed. Domain sub-scores were summed to yield a total raw score. This was divided by the total possible score and multiplied by 100 to produce the final score. Each subscale score can be calculated in the similar approach.
Time Frame: Baseline (Visit 2), Week 6 (Visit 3), Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 93
Scores on a scale
  Baseline (Visit 2) | 58.3 (26.48)
  Week 6 (Visit 3) | 58.4 (24.93)
  Week 12/ET (Visit 4) | 57.2 (25.53)
  Week 12 LOCF (Study Endpoint) | 57.2 (25.39)

10. Secondary Outcome: Change From Baseline in DAD Total Score by Visit
Description: as for outcome 9
Time Frame: Baselinw, Week 6 (Visit 3) and Week 12 (Visit 4) or ET Visit, Week 12 LOCF (Study Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil Hydrochloride (HCl)
Number analyzed (Participants) | 93
Scores on a scale
  Baseline | 58.3 (26.48)
  Change from Baseline at Week 6 (Visit 2) | -1.1 (8.52)
  Change from Baseline at Week 12/ET (Visit 4) | -1.1 (14.38)
  Change from Baseline at Week 12 LOCF | -1.1 (14.30)
Statistical Analysis 1: Comparison: Donepezil Hydrochloride (HCl); Week 6 (Visit 3); Test type: Superiority or Other; p = 0.2327, t-test, 2 sided — Significance level of 0.05
Statistical Analysis 2: Comparison: Donepezil Hydrochloride (HCl); Week 12/ET (Visit 4); Test type: Superiority or Other; p = 0.4724, t-test, 2 sided — Significance level of 0.05
Statistical Analysis 3: Comparison: Donepezil Hydrochloride (HCl); Week 12 LOCF - Study Endpoint; Test type: Superiority or Other; p = 0.4724, t-test, 2 sided — Significance level of 0.05

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) and serious adverse events (SAEs) were collected from Screening Visit 1 (-21 to -14 days) until Week 12 Visit 4 (Day 84) or early termination. AEs/SAEs were collected for approximately 4 months.
Description: Treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events were reported. TEAEs were defined as events that occurred after the first dose of study drug or a pre-existing condition that worsened after starting study drug. The safety population was analyzed and included enrolled participants who received at least one dose of study drug.
Arm/Group | Donepezil Hydrochloride (HCl)
All-Cause Mortality (participants affected / at risk) | 2/97
Serious Adverse Events (participants affected / at risk) | 12/97
Other Adverse Events (participants affected / at risk) | 56/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Hydrochloride (HCl) (N=97)
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastric volvulus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Muscle mass (Musculoskeletal and connective tissue disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Alcohol abuse (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Hydrochloride (HCl) (N=97)
Nausea (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Urinary tract infection (Infections and infestations) | 4
Vomiting (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Depression (Psychiatric disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Irritability (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 2
Oedema peripheral (General disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 2
Weight decreased (Investigations) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other